CLINICAL TRIAL: NCT05273242
Title: WHO Solidarity Trial Plus: An International Randomised Trial of Additional Treatments for COVID-19 in Hospitalised Patients Who Are All Receiving the Local Standard of Care in Nepal
Brief Title: Add-on Study on WHO Solidarity Trial Plus for COVID-19 in Nepal
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nepal Health Research Council (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Dr. Pradip Gyanwali,MD, Executive Chief (Member Secretary), Nepal Health Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Solidarity Trial Plus In Nepal; ISRCTN18066414 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2021-12-10; First posted 2022-03-10 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Artesunate

STUDY DESIGN:
Intervention Model Description: Same as that of WHO solidarity Trial Plus , Please refer to the ISRCTN18066414
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Artesunate (Experimental): Please refer to the WHO solidarity Trial Plus Protocol ISRCTN18066414
  Interventions: Drug: Artesunate Injection
- Imatinib (Experimental): Please refer to the WHO solidarity Trial Plus Protocol ISRCTN18066414
  Interventions: Drug: Artesunate Injection
- Infliximab (Experimental): Please refer to the WHO solidarity Trial Plus Protocol ISRCTN18066414
  Interventions: Drug: Artesunate Injection
- Local Standard of Care (No Intervention): No other Intervention Given except the local standard of care

INTERVENTIONS:
Drug: Artesunate Injection — * Artesunate: 2.4 mg/kg/dose at 0 hours, 12 hours, and 24 hours and thereafter every 24 hours; IV injection; duration of treatment 7 days. This is the standard dose recommended for the treatment of severe malaria.
  * Infliximab: 5 mg/kg/dose (once only), single IV infusion over 2 hours. This is the standard dose that is given repeatedly for the treatment of psoriasis.
  * Imatinib: 400 mg/dose; orally once daily; duration of treatment 14 days. This is the standard maintenance dose which is at the lower end of that used for several years in the treatment of hematological malignancies.
  Other Names: Imatinib. Infliximab
  Arms: Artesunate; Imatinib; Infliximab

SUMMARY:
Proposal for Sub-Study to be conducted with the WHO Solidarity Plus Trial:

Apart from the data been collected as per the WHO Solidarity Trial Plus protocol, Nepal Health Research Council will conduct a sub-study to evaluate some components which are felt to be important in the local context but have not been included as part of the Solidarity Trial Plus. Rather that conducting a separate study, the following components can be evaluated by collecting additional data as a part of sub-study in the local context.

DETAILED DESCRIPTION:
Patients enrolled in the WHO Solidarity Plus trial will also be consented for this sub-study for further data collection in the following four categories. No additional tests or investigations will be performed.

1. Socio-economic factors: Investigators have added the socio-demographic factors in our data collection tool to get insight into the socio-demographic distribution of the hospitalized patients enrolled in the study. These data will help to understand the disease distribution in the local context. These factors are listed in the table below.
2. Laboratory investigations: There is no provision to collect the information on investigations including laboratory tests and radiological findings in the current WHO Solidarity protocol. These data will help to analyze the systemic effects of the study drugs and help to verify AEs/SAEs/SUSARs reported by the investigators. Hence, Investigators have added the information related to the various investigations in our study. Investigators will not collect additional bio samples or conduct any additional laboratory or radiological investigations. However, if such information is available, Investigators will collect such data and record the information in our local study database.
3. Immunization status: Investigators currently do not have studies looking at impact of vaccines on hospitalization, severity and mortality in Nepal. Data related to the vaccination status is not included in the Solidarity protocol. After the availability of the vaccine, vaccination status may be a confounding factor to determine the mortality outcome. Hence, investigators plan to add vaccine status as one of the variables in the sub-study.
4. Follow up after discharge: Investigators plan to add follow up visit or phone calls after the discharge which is not included in the current WHO Solidarity protocol. The study team will conduct follow up visits or phone calls each week to assess the status of the patients until 28 days and each month for six months thereafter from the date of first randomization. The follow up visits will be done by telephone call either to the patient or the patient's relative. Study team will ask about the condition of the patient since the time of discharge and find out general health status (normal versus abnormal), re-hospitalization, and mortality

ELIGIBILITY:
Inclusion Criteria:

* Recently hospitalized (or already in hospital) with laboratory-confirmed COVID
* In the view of their doctors, no contra-indication to any potentially relevant study drug.
* Voluntary Participation

Exclusion Criteria:

* In the view of the randomising doctor, ANY of the AVAILABLE study drugs are contra-indicated (eg, because of patient characteristics, chronic liver or heart disease, or some concurrent medication).
* If expected to be transferred within 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Hospital Mortality | The duration in the number of days calculated from the first date of randomization of the patient till the final outcome in the hospital that the first documented progression or death due to COVID 19 up to 28 days whichever comes first
  To assess the incidence of hospital mortality in the patient who are receiving study drug in addition to local standard of care

SECONDARY OUTCOMES:
Assessment of duration of hospital stay, | The duration in the number of days calculated from the first date hospitalization due to COVID 19 until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 28 days
  To assess the number of days in hospital due to COVID 19 in the patient who are receiving study drug in addition to local standard of care
Initiation of ventilation | The number of days calculated from date of randomization until the date of initiation of ventilation, assessed up to 28 days
  To asses number of days ventilation requirement in the patient who are receiving study drug in addition to local standard of care
Assessment of Serious adverse reactions (SAE) | Number of Serious Adverse Effect (SAE) calculated from the day of randomization upto 28 days
  To assess the incidence of any Serious adverse reactions (SAE) in the patient who are receiving study drug in addition to local standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marie-Pierre Preziosi, Study Director — WHO Solidarity Trial Plus
Locations (5):
- Nepal (5):
  - Chitwan Medical College, Bharatpur, Bagmati
  - Civil Service Hospital, Kathmandu, Bagmati
  - Patan Academy of Health Sciences, Lalitpur, Bagmati
  - Lumbini Provincial Hospital, Butwāl, Lumbini
  - Narayani Hospital, Birgunj, Madhesh

IPD SHARING:
Plan to Share IPD: No